CLINICAL TRIAL: NCT06976385
Title: Clinical Impact of White Tea and Wheat Grass on Color Enhancement of White Spot Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mariam Mohamed Taha Elnems, Lecturer of conservative dentistry, NewGiza University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-CL-23-14b
Record Dates: First submitted 2025-05-09; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: White Spot Lesions [Initial Caries] on Smooth Surface of Tooth

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- White tea (Experimental): Participants prepared white tea mouth rinse to rinse thoroughly . At each rinsing, 10 mL of the solution was swished around the mouth for about 60 s and then spited This procedure was performed twice per day for 1 , and 3 months
  Interventions: Dietary Supplement: White tea
- Wheat grass solution (Experimental): Participants prepared wheat grass solution mouth rinse to rinse thoroughly . At each rinsing, 10 mL of the solution was swished around the mouth for about 60 s and then spited This procedure was performed twice per day for 1 , and 3 months
  Interventions: Dietary Supplement: Wheat grass solution

INTERVENTIONS:
Dietary Supplement: White tea — White tea mouth rinse applied topically twice daily.
  Arms: White tea
Dietary Supplement: Wheat grass solution — wheat grass solution mouth rinse applied topically twice daily.
  Arms: Wheat grass solution

SUMMARY:
The current study aimed to evaluate the color change potential of wheat grass and white tea on post orthodontic white spot lesions (WSLs). Materials and Methods: A total of 12 patients were divided into two main groups A1 and A2 according to type of treatment agent (n=6). The A1 group used 10% white tea solution while the A2 group used 10% wheat grass solution. Shade evaluation was conducted using VITA Easyshade V spectrophotometer. Baseline L a b values of WSLs were detected right after orthodontic bracket removal. Patients were requested to rinse with the treatment agent for 1 minute, twice per day. The mean L,a,b values were recorded after 1 month and after 3 months . ΔE values were calculated between baseline, 1 month and 3 months after the treatment agent application and subjected to statistical analysis using one way ANOVA with p>0.05. Also, Standardized photographs were taken at baseline, after 1 and 3 months. Each WSL was photographed twice with the 1st photograph taken of wet teeth and the 2nd one after prolonged air-drying in order to perform ICDAS II scoring.

ELIGIBILITY:
Inclusion Criteria:

1. Age range between 15-18 years.
2. Good oral hygiene
3. Obvious area of WSL was found around the fixed orthodontic brackets.
4. Included teeth should be free of any restorations

Exclusion Criteria:

- : 1. Cavitated enamel surface. 2. Presence of any restorations including the labial surface of the involved teeth.

3. Presence of any environmental or developmental enamel defect such as enamel hypoplasia, fluorosis, stains, and trauma sites on teeth before orthodontic treatment. 4. Allergy to tea and/or wheat

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
ΔE values were calculated | after 1 month and after 3 months
  The mean L,a,b values were recorded . ΔE values were calculated

CONTACTS AND LOCATIONS:
Locations (1):
- Al Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No